CLINICAL TRIAL: NCT04031651
Title: Key Specialized Monitoring of Clinical Safety of Pudilan Xiaoyan Oral Liquid in the Real World
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: China Academy of Chinese Medical Sciences (Other)
Collaborators: Xiyuan Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Yanming Xie, Deputy Director, China Academy of Chinese Medical Sciences
Other Study IDs: PUDILAN
Record Dates: First submitted 2019-07-12; First posted 2019-07-24 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-06

CONDITIONS: Respiratory Infectious Diseases
Keywords: Pudilan Xiaoyan Oral Liquid; Safety monitoring
MeSH Terms: interventions — Pudilan xiaoyan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Pudilan Xiaoyan Oral Liquid — In the respiratory and emergency departments of the hospitals under surveillance, the medication of Pudilan Xiaoyan Oral Liquid is observed for those aged 18-80 years who strictly follow the prescription of the instructions.

SUMMARY:
To obtain the characteristics of adverse reactions/incidents, analyze the influencing factors and calculate the incidence of adverse reactions/incidents monitored by Pudilan Xiaoyan Oral Liquid in key specialties in the real world, so as to provide a basis for clinical safe and rational drug use.

ELIGIBILITY:
Inclusion Criteria:

* (1)Upper respiratory tract infection patients using Pudilan antiphlogistic oral liquid ;
* (2)Aged between 18 and 80.

Exclusion Criteria:

* Lactating women, pregnant women, pregnant planners, psychiatric patients, etc.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: To obtain the characteristics of adverse reactions/incidents, analyze the influencing factors and calculate the incidence of adverse reactions/incidents monitored by Pudilan Xiaoyan Oral Liquid in key specialties in the real world, so as to provide a basis for clinical safe and rational drug use.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2019-07-17 (Estimated); Primary Completion 2019-07-17 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Drug Reaction | 7 days
  Incidence of Reduning Injection'Adverse Drug Reaction（ADRs）and Identify Factors That Contributed to the Occurrence of the Adverse Drug Reaction

SECONDARY OUTCOMES:
The Ratio of Body Temperature to Normal | 7 days
  The Ratio of Body Temperature to Normal(Lower Than 37.3ºC)
Change of liver function | 7 days
  Observation of liver function in at least 3000 patients before and after medication.The liver function includes glutamic-pyruvic transaminase,glutamic-oxalacetic transaminase.To observe whether the above liver function indexes appear abnormal once after medication.
Change of renal function | 7 days
  Observation of renal function in at least 3000 patients before and after medication.The renal function includes creatinine,usea nitrogen.To observe whether the above renal function indexes appear abnormal once after medication.

CONTACTS AND LOCATIONS:
Overall Officials: Yanming Xie, BA, Principal Investigator — Institute of Basic Research in Clinical Medicine, China Academy of Chinese

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang M, Wang L, Liu F, Chen R, Wang Z, Cui X, Li Y, Xie Y. Clinical Safety of Pudilan Xiaoyan Oral Liquid for the Treatment of Upper Respiratory Tract Infection in the Real World: Protocol for a Prospective, Observational, Registry Study. JMIR Res Protoc. 2025 Mar 21;14:e65789. doi: 10.2196/65789. PMID 40117581